CLINICAL TRIAL: NCT02132312
Title: A Randomized, Double-Masked, Parallel-Group, Phenylephrine-Controlled Study of the Effect of OMS302 Added to Standard Irrigation Solution on Intraoperative Pupil Diameter and Acute Postoperative Pain in Children Ages Birth Through Three Years Undergoing Unilateral Cataract Extraction With or Without Lens Replacement
Brief Title: A Randomized Study in Children Ages Birth Through Three Years Undergoing Unilateral Cataract Extraction With or Without Lens Replacement
Acronym: ILR7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMS302-ILR-007
Record Dates: First submitted 2014-05-01; First posted 2014-05-07 (Estimated); Results first posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Unilateral Cataract Extraction; Congenital Cataract
Keywords: Cataract; Lens replacement; pediatric
MeSH Terms: conditions — Cataract | interventions — Oxymetazoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OMS302 (Experimental): OMS302 diluted in balanced salt solution (BSS) and administered as irrigation solution
  Interventions: Drug: OMS302
- Phenylephrine HCl (Active Comparator): Phenylephrine diluted in balanced salt solution (BSS) and administered as irrigation solution
  Interventions: Drug: Phenylephrine HCl

INTERVENTIONS:
Drug: OMS302
  Arms: OMS302
Drug: Phenylephrine HCl
  Arms: Phenylephrine HCl

SUMMARY:
The purpose of this study is to evaluate the effect of OMS302 compared to phenylephrine when administered in irrigation solution during cataract extraction on intraoperative pupil diameter, acute postoperative pain, and safety in children birth through 3 years.

DETAILED DESCRIPTION:
This study is a randomized, parallel-group, double-masked, phenylephrine-controlled study of OMS302 in young children ages birth through three years undergoing unilateral cataract extraction with or without lens replacement. Administration of test irrigation solutions will take place in a double-masked fashion.

Intraoperative pupil size will be determined by measurement of pupil diameter from still photos captured from video recordings of the procedure. Pupil diameter measurements will be performed immediately prior to the initial incision and at one-minute intervals until the end of the procedure (wound closure). Pain will be assessed by the Alder Hey Triage Pain Score.

ELIGIBILITY:
Inclusion Criteria:

1. Are 0 through three years of age at the time of surgery.
2. Are to undergo unilateral primary cataract extraction with or without lens replacement.
3. Have informed consent and Health Insurance Portability and Accountability Act (HIPAA) Authorization provided by a parent or legal guardian in accordance with local regulations and governing IRB/IEC requirements prior to any procedures or evaluations performed specifically for the sole purpose of this study.
4. A parent or legal guardian has indicated that they understand and are able, willing, and likely to fully comply with study procedures and restrictions.

Exclusion Criteria:

1. Corneal diameter less than nine millimeters in the study eye.
2. Hypersensitivity to phenylephrine, ketorolac, or other NSAIDs, including aspirin, or latex.
3. Surgeon's expectation that the protocol-specified mydriatic regimen will not be adequate to perform the procedure and that additional mydriatic treatment (pharmacological or mechanical) will be required.
4. Presence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, endocrine, neurological, psychiatric, respiratory, or other medical condition that could increase the risk to the subject as determined by the Investigator.
5. Presence of active or suspected viral, bacterial, or fungal disease in the study eye.
6. Use of any topical medication in the study eye within seven days prior to surgery, except for medications needed to examine the eye or prepare for surgery.
7. Have a post-traumatic cataract.
8. History of uveitis or evidence of past uveitis such as synechiae or keratic precipitates in the study eye.
9. Have an ocular neoplasm in the study eye.
10. Have a clinically significant infection.
11. Have suspected permanent or low vision in the fellow non-study eye, unless caused by a cataract. The study eye must not be the subject's only good eye.
12. Use of systemic corticosteroids or NSAIDs in the seven days prior to surgery.
13. Have a history of clinically significant corticosteroid-induced intraocular pressure increase.
14. Use of any medication for ocular hypertension or glaucoma in the study eye.
15. Use of monoamine oxidase inhibitors for 21 days preoperatively.
16. Prior participation in a clinical study of OMS302.
17. Participating in any investigational drug or device trial within the 30 days prior to the day of surgery.
18. History of intraocular non-laser surgery in the study eye within the three months prior to the day of surgery, or intraocular laser surgery in the study eye within 30 days prior to the day of surgery.
19. Presence of any condition that the Investigator believes would put the subject at risk or confound the interpretation of the study data.
20. Be a member of the immediate family of the Investigator or employees of the investigative site. Immediate family is defined as the Investigator's or employees' natural or legally adopted child (including a stepchild living in the Investigator's household), or grandchild.

Ages: 1 Day to 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09-12 (Actual); Study Completion 2016-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Whitaker, MD, Study Director — Omeros Corporation
Locations (11):
- United States (11):
  - Los Angeles, California
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Boston, Massachusetts
  - Detroit, Michigan
  - Charleston, North Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Madison, Wisconsin

REFERENCES:
- [Background] Wilson ME, Trivedi RH, Plager DA. Safety and efficacy data supporting U.S. FDA approval of intracameral phenylephrine and ketorolac 1.0%/0.3% for pediatric cataract surgery: clinical safety and pupil and pain management. J Cataract Refract Surg. 2020 Jun;46(6):873-878. doi: 10.1097/j.jcrs.0000000000000194. PMID 32221151

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 78 participants enrolled in the study. 6 participants were consented and randomized but did not receive OMS302 or Phenylephrine HCl. Out of the 72 participants who received OMS302 or Phenylephrine HCl, 3 participants did not complete the study. One participant was randomized to OMS302, but received Phenylephrine HCl. This participant was included in the OMS302 group in baseline analyses and in the Phenylephrine HCl group in safety analyses.
Groups:
- OMS302: OMS302 diluted in balanced salt solution (BSS) and administered as irrigation solution
  OMS302
- Phenylephrine HCl: Phenylephrine diluted in balanced salt solution (BSS) and administered as irrigation solution
  Phenylephrine HCl
Period: Overall Study
Arm/Group | OMS302 | Phenylephrine HCl
Started | 37 | 41
Completed | 31 | 38
Not Completed | 6 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: 78 participants enrolled in the study. 6 participants were consented and randomized but did not receive OMS302 or Phenylephrine HCl. One out of 72 participants was randomized to OMS302 but received Phenylephrine HCl. This participant was included in the OMS302 group in baseline analyses and in the Phenylephrine HCl group in safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | OMS302 | Phenylephrine HCl | Total
Number analyzed (Participants) | 33 | 39 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.0 (1.1) | 1.4 (1.2) | 1.2 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 17 | 20 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 10 | 10
  Not Hispanic or Latino | 33 | 29 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 26 | 30 | 56
  More than one race | 1 | 6 | 7
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Pupil Diameter
Description: Mean Area-under-the-Curve (AUC) Analysis of Change From Baseline in Pupil Diameter (mm/min) During Surgery Excluding Subjects with In-evaluable Videos.
Time Frame: From surgery baseline (pre-incision) through surgery end (time of cortical clean-up/wound closure), the mean time of surgery duration is 35.46 minutes with a standard deviation of 19.98.
Population: There were 61 evaluable videos, one for each subject.
Measure: Mean (Standard Deviation); unit: millimeters*minutes
Arm/Group | OMS302 | Phenylephrine HCl
Number analyzed (Participants) | 30 | 31
millimeters*minutes | 0.14 (0.474) | 0.20 (0.600)

2. Primary Outcome: Acute Postoperative Pain
Description: Mean AUC Analysis of Postoperative pain as measured using the Alder Hey Triage Pain Score at 3, 6, 9, and 24 hours after surgery. The primary analysis of Alder Hey Triage Pain Score was similar to the primary analysis of the change in pupil diameter using AUC. The Alder Hey Triage Pain Score identifies five categories of observations: voice/cry, facial expression, posture, movement, and color. Each of these has a possible score of 0, 1, or 2, resulting in a total score ranging between 0 and 10. A total score of zero means the subject experienced no pain, as the 5 categories added up totals zero. A total score of 10 means the subject experienced a lot of pain and is the worst possible outcome, as the 5 categories added up totals 10.
  Parent responses in a diary with a score of 0, 1, or 2.
  1. Cry or voice, 0=no compliant/cry, 1=Consolable, 2=Inconsolable
  2. Facial Expression, 0=Normal, 1=Short grimace <50% of time, 2=Long grimace >50% of time
  3. Posture, 0=Normal, 1=Touching/rub
Time Frame: 24 hours
Population: There were 71 participants with evaluable postoperative pain scores.
Measure: Mean (Standard Deviation); unit: score*hours
Arm/Group | OMS302 | Phenylephrine HCl
Number analyzed (Participants) | 33 | 38
score*hours | 0.44 (0.742) | 0.65 (0.943)

3. Primary Outcome: Safety as Measured by Treatment-emergent Adverse Events, the Number of Affected Patients/at Risk (%) and the Number of Events.
Description: Safety as assessed by the incidence of adverse events and serious adverse events up until the last visit at Day 90.
Time Frame: 90 days
Population: 78 participants enrolled in the study. 6 participants were consented and randomized but did not receive OMS302 or Phenylephrine HCl. Safety analyses were based on the safety population. Out of the 72 participants, one participant was randomized to OMS302 but received Phenylephrine HCl. This participant was included in the Phenylephrine HCl group for safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | OMS302 | Phenylephrine HCl
Number analyzed (Participants) | 32 | 40
Participants | 15 | 18

ADVERSE EVENTS:
Time Frame: 90 days
Description: 78 participants enrolled in the study. 6 participants were consented and randomized but did not receive OMS302 or Phenylephrine HCl. Safety analyses were based on the safety population. One out of 72 participants was randomized to OMS302 but received Phenylephrine HCl. This participant was included in the Phenylephrine HCl group for safety analyses.
Arm/Group | OMS302 | Phenylephrine HCl
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/40
Serious Adverse Events (participants affected / at risk) | 2/32 | 0/40
Other Adverse Events (participants affected / at risk) | 15/32 | 18/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OMS302 (N=32) | Phenylephrine HCl (N=40)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OMS302 (N=32) | Phenylephrine HCl (N=40)
Persistent Pupillary Membrane (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Acquired Epiblepharon (Eye disorders) | 0 (0) | 1 (1)
Anisometropia (Eye disorders) | 0 (0) | 1 (1)
Anterior Capsule Contraction (Eye disorders) | 0 (0) | 1 (1)
Anterior Chamber Inflammation (Eye disorders) | 1 (1) | 0 (0)
Anterior Chamber Opacity (Eye disorders) | 2 (2) | 2 (2)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 3 (3)
Conjunctival Hyperaemia (Eye disorders) | 1 (1) | 1 (1)
Dry Eye (Eye disorders) | 1 (1) | 0 (0)
Eyelid Ptosis (Eye disorders) | 1 (1) | 0 (0)
Iris Adhesions (Eye disorders) | 1 (1) | 0 (0)
Retinal Haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Vitreous Fibrin (Eye disorders) | 1 (1) | 0 (0)
Vitreous Haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Immunisation Reaction (Immune system disorders) | 0 (0) | 2 (2)
Bronchiolitis (Infections and infestations) | 2 (2) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Corneal Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraocular Pressure Increased (Investigations) | 2 (2) | 2 (2)
Vesicoureteric Reflux (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eustacian Tube Operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes